CLINICAL TRIAL: NCT07139119
Title: Impact of a Health Belief Model-Based Educational Intervention on Skin Cancer Protective Behaviors Among Female Healthcare Workers
Brief Title: Educational Intervention on Skin Cancer Protective Behaviors Among Female Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arash Salahshouri, Faculty member, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IR.AJUMS.REC.1401.129
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Promoting Skin Cancer Protective Behaviors
Keywords: Educational intervention; Health Belief Model; Cancer; Skin cancer; Healthcare Workers
MeSH Terms: conditions — Neoplasms; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group quasi-experimental design, where female healthcare workers are assigned to either an intervention group or a comparison group. Both groups were followed concurrently over a two-month period. The intervention group received a multicomponent blended educational program based on the Health Belief Model (HBM), delivered through face-to-face sessions and WhatsApp messaging. The comparison group did not receive any educational intervention. Outcomes related to skin cancer knowledge, Health Belief Model constructs, and protective behaviors against ultraviolet radiation were measured and compared at baseline and two months post-intervention. This design allows a direct evaluation of the intervention's effectiveness compared to usual conditions without educational input.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention Group (Experimental): Female healthcare workers participated in a multilevel educational intervention based on the Health Belief Model (HBM) to enhance skin cancer protective behaviors. The program consisted of seven 45-minute sessions delivered both face-to-face and virtually via WhatsApp. The sessions focused on improving knowledge and modifying HBM construct. Educational materials included pamphlets, video clips, group discussions, and motivational messages. Reminders and posters were used in the workplace to reinforce learning and encourage sustained behavior change.
  Interventions: Behavioral: Health Belief Model-Based Educational Program for Skin Cancer Prevention Among Female Healthcare Workers
- Arm 2: Control Group (No Intervention): Participants in the control group did not receive any educational intervention during the study period. They continued with their usual work routine and standard health education programs available at their workplaces. Assessments of their knowledge, health beliefs, and protective behaviors related to skin cancer were conducted at baseline and two months later to serve as a comparison for evaluating the effectiveness of the intervention.

INTERVENTIONS:
Behavioral: Health Belief Model-Based Educational Program for Skin Cancer Prevention Among Female Healthcare Workers — This blended educational intervention employs the Health Belief Model (HBM) to promote skin cancer preventive behaviors in female healthcare workers in Ahvaz, Iran. The 7-session program (each 45 minutes) combines in-person training with WhatsApp-based follow-ups.
  Participant Components:
  * Structured sessions targeting knowledge and HBM constructs such as perceived susceptibility, severity, benefits, barriers, self-efficacy, and cues to action.
  * Use of multimedia tools including videos, pamphlets, and interactive discussions.
  * Motivational messaging, stress management clips, and role-modeling techniques to build self-efficacy.
  * Visual cues such as posters placed in healthcare workplaces.
  * Daily reminder messages to reinforce behavior change.
  Unique aspects distinguishing this intervention include its specific tailoring for female healthcare workers in a high UV-exposure region, the combined digital and face-to-face delivery approach, and comprehensive focus on all HBM construc
  Arms: Arm 1: Intervention Group

SUMMARY:
The goal of this clinical trial is to assess whether an educational intervention based on the Health Belief Model (HBM) can effectively improve skin cancer protective behaviors, knowledge, and related health beliefs among female healthcare workers in Ahvaz, Iran. The main questions it aims to answer are:

* Does the HBM-based educational program increase participants' knowledge about skin cancer, its risk factors, and preventive measures?
* Does the intervention improve key HBM constructs such as perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy, and cues to action, leading to enhanced protective behaviors against skin cancer?

Researchers will compare an intervention group receiving a multicomponent educational program-including seven 45-minute sessions delivered both in-person and via WhatsApp-tailored to HBM constructs, with a comparison group receiving no intervention, to determine the intervention's effectiveness.

Participants will:

* Attend structured educational sessions covering skin cancer symptoms, risks, prevention strategies, behavioral barriers, motivation, and self-efficacy enhancement, using multimedia tools and group discussions
* Receive reminder messages and educational materials to facilitate behavior change
* Complete validated questionnaires assessing knowledge, HBM constructs, and protective behaviors before the intervention and two months afterwards

This study will evaluate if implementing a theory-driven, blended educational intervention can successfully promote protective behaviors and health beliefs related to skin cancer prevention among female healthcare workers.

DETAILED DESCRIPTION:
This clinical trial study was conducted from 2022 to 2023 in health centers of Ahvaz, Iran, to evaluate the effectiveness of an educational intervention based on the Health Belief Model (HBM) in promoting skin cancer protective behaviors among female healthcare workers (HCWs). The study employed a two-group parallel design, randomly allocating 160 participants into an intervention group (n=54) and a comparison group (n=106). Eligible participants included female HCWs employed in the selected centers, with smartphone access and the ability to engage with digital educational content.

The educational program was developed according to HBM constructs, including perceived susceptibility, perceived severity, perceived benefits, perceived barriers, cues to action, and self-efficacy. The intervention consisted of seven 45-minute sessions delivered over two months using a blended approach combining in-person workshops and WhatsApp-based virtual education. Teaching methods included lectures, multimedia presentations, group discussions, motivational messaging, and reminder posters strategically placed in the workplace.

The content was tailored based on baseline knowledge and behavioral assessments. Early sessions addressed skin cancer symptoms, risk factors, and complications to raise awareness and perceived risk. Subsequent sessions emphasized the advantages of protective behaviors, addressed and sought to reduce perceived barriers, and incorporated stress management and motivational techniques to enhance self-efficacy.

Data collection employed a validated researcher-designed questionnaire covering demographic variables, knowledge about skin cancer, HBM constructs, and adherence to UV protective behaviors. Assessments were performed at baseline and two months post-intervention.

Statistical analyses included descriptive statistics, Chi-square tests for categorical variables, and independent and paired t-tests to compare continuous variables within and between groups. Analysis of covariance (ANCOVA) controlled for confounding factors when evaluating intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Employment at Ahvaz healthcare centers,
* Absence of specific dermatological conditions,
* Provision of informed consent,
* Having a smartphone and knowing how to use it, and
* Non-participation in concurrent similar educational interventions.

Exclusion Criteria:

* Absence from more than two training sessions,
* Physical limitations preventing further participation,
* Incomplete or invalid questionnaire .

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Changes in Skin Cancer Protective Behaviors | Baseline (pre-intervention) and 2 months post-intervention.
  Skin cancer protective behaviors among female healthcare workers were assessed using a validated, researcher-developed questionnaire. The instrument included multiple items evaluating behaviors such as applying sunscreen, wearing protective clothing (wide-brimmed hats, long-sleeved shirts, gloves), and using sunglasses. Responses were measured on a 5-point Likert scale ranging from 1 ("Never") to 5 ("Always"). Protective behaviors were expressed as the average score across items, with higher scores indicating more frequent and consistent engagement in skin cancer prevention practices.

SECONDARY OUTCOMES:
Changes in Cognitive-Behavioral Constructs Related to Skin Cancer Prevention | Before and two months after the intervention
  This outcome assesses changes in Health Belief Model (HBM)-based constructs related to skin cancer prevention, including perceived susceptibility (5 items; score range: 5-25), perceived severity (6 items; score range: 6-30), perceived benefits (5 items; score range: 5-25), perceived barriers (6 items; score range: 6-30), cues to action (4 items; score range: 4-20), self-efficacy (7 items; score range: 7-35), and knowledge (15 items; score range: 0-15). All constructs except perceived barriers were scored on a 5-point Likert scale ranging from "Strongly Agree" (score 5) to "Strongly Disagree" (score 1), where higher scores indicate more favorable outcomes such as greater perceived susceptibility, severity, benefits, self-efficacy, and cues to action. Items related to perceived barriers were reverse scored, so that higher scores indicate fewer perceived barriers. These constructs were measured using validated, researcher-developed questionnaires at baseline and two months after the inte

CONTACTS AND LOCATIONS:
Overall Officials: Arash Salahshouri, Ph.D., Principal Investigator — Ahvaz Jundishapur University of Medical Sciences
Locations (1):
- Ahwaz West Health Center, Ahvāz, Khouzestan, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Public release of these data is not part of the research plan. However, upon reasonable request from researchers, and with ethics committee approval and strict confidentiality maintained, participant data can be shared with researchers in a controlled and limited manner.